CLINICAL TRIAL: NCT05582707
Title: A Non-Randomized Controlled Trial to Examine the Safety and Suitability of Supplementing Early Minimally Invasive Parafascicular Surgery (MIPS) for Clot Evacuation of Basal Ganglia Intracerebral Hemorrhage (ICH) With Pioglitazone
Brief Title: Safety and Suitability of Supplementing Early MIP Surgery (MIPS) of ICH With Pioglitazone
Acronym: ENRICHPLUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of Financial Sponsor
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Nico Corporation (Industry)
Responsible Party: Principal Investigator, Marc Simard, Principal Investigator, Clinical Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00102344
Record Dates: First submitted 2022-10-03; First posted 2022-10-17 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Intracerebral Haemorrhage, Intraventricular
Keywords: Pioglitazone; Basal Ganglia Intracerebral Hemorrhage (ICH); Minimally Invasive Parafascicular Surgery
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: All subjects enrolled in this trial will be in the Experimental arm and receive intervention of MIPS + Pioglitazone. These patients will be compared to a dataset of subjects who have already undergone MIPS alone in a previous trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MIPS + Pioglitazone (Experimental): 20 Subjects will undergo MIPS for evacuation of ICH using the BrainPath access device plus perioperative pioglitazone for 3 weeks
  Interventions: Drug: Pioglitazone 15mg
- MIPS Alone (No Intervention): This trial will compare it's subjects to subjects who have previously undergone MIPS for evacuation of ICH using the BrainPath access device as part of the ENRICH trial (NCT02880878). These subjects will be enrolled at an ENRICH trial site independent of our Institution. Deidentified patient information from 20 subjects in this group, who will be matched to those in the ENRICH-PLUS group, will be provided to the principal investigator for comparison of outcomes.

INTERVENTIONS:
Drug: Pioglitazone 15mg — Study participants will be administered pioglitazone (15 mg tablet) either p.o. or enteral (via nasogastric tube). The first dose may be administered prior to surgery or within 3 hours of the end of surgery but must be administered within 24 hours of the index event or time last known normal (TLKN). Pioglitazone (15 mg tablet) administration will continue 3 times daily for 3 weeks, including after hospital discharge, if applicable.
  Arms: MIPS + Pioglitazone

SUMMARY:
This is an exploratory single-center prospective study of 20 subjects with primary basal ganglia ICH who will receive early MIPS in combination with perioperative pioglitazone treatment. Outcomes will be compared to matched subjects with basal ganglia ICH who undergo MIPS alone as part of the ENRICH trial. This study will take approximately two years to complete.

DETAILED DESCRIPTION:
Study Arms:

Group 1: 20 Subjects will undergo MIPS for evacuation of ICH using the BrainPath access device plus perioperative pioglitazone for 3 weeks

Group 2: Subjects will undergo MIPS for evacuation of ICH using the BrainPath access device as part of the ENRICH trial (NCT02880878). These subjects will be enrolled at an ENRICH trial site independent of our Institution. Deidentified patient information from 20 subjects in this group, who will be matched to those in the ENRICH-PLUS group, will be provided to the principal investigator for comparison of outcomes.

Consent for study participation will be obtained from the patient or the LAR only after fulfilling all inclusion and exclusion criteria either before or after MIPS, which will be scheduled as a standard institutional procedure outside the realm of the study.

Study participants will be administered pioglitazone (15 mg tablet) either p.o. or enteral (via nasogastric tube). The first dose may be administered prior to surgery or within 3 hours of the end of surgery but must be administered within 24 hours of the index event or time last known normal (TLKN). Pioglitazone (15 mg tablet) administration will continue 3 times daily for 3 weeks, including after hospital discharge, if applicable.

Following completion of pioglitazone, subjects will be followed at days 30, 90, 120 and 180 post MIPS. In addition to AE monitoring during these follow up's, a utility-weighted mRS (uw-mRS) at 180 days will serve as the primary end point.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. CT scan demonstrating an acute, spontaneous, primary basal ganglia ICH
3. ICH volume between 30 - 80 mL as calculated by the ABC/2 method
4. Study intervention can reasonably be initiated within 24 hours after the onset of stroke symptoms. In situations with unclear time of onset, then the onset will be considered the time that the subject was last known to be well
5. Glasgow Coma Score (GCS) 5 - 14
6. Historical Modified Rankin Score 0 or 1
7. Consent by patient or LAR to MIS evacuation of the ICH based on best medical practice1
8. Time to pioglitazone treatment ≤ 24 hours from symptom onset or TLKN1

Exclusion Criteria:

1. Ruptured aneurysm, arteriovenous malformation (AVM), vascular anomaly, moyamoya disease, hemorrhagic conversion of an ischemic infarct, or bleeding into a known neoplastic lesion
2. NIHSS< 5, bilateral fixed dilated pupils, extensor motor posturing, unstable mass or evolving intracranial compartment syndrome
3. Intraventricular extension of the hemorrhage estimated to involve >50% of either of the lateral ventricles (External ventricular drain (EVD) to treat intracranial pressure (ICP) or hydrocephalus is allowed)
4. Primary thalamic ICH or infratentorial intraparenchymal hemorrhage including midbrain, pons or cerebellum
5. Evidence of active bleeding involving a retroperitoneal, gastrointestinal, genitourinary, or respiratory tract site
6. Severe kidney or liver disease (serum ALT > 2.5 x ULN) with active coagulopathy
7. Patients requiring long-term anticoagulation that needs to be initiated < 5 days from index ICH; patient must not require Coumadin (anticoagulation) during the first 30 days (reversal of anticoagulation is permitted for medically stable patients who can safely tolerate the short-term risk of reversal)
8. Use of anticoagulants that cannot be rapidly reversed, uncorrected coagulopathy or known clotting disorder
9. Platelet count < 75,000
10. International Normalized Ratio (INR) > 1.4 after correction or inability to sustain INR ≤ 1.4 using short- and long-active procoagulants (such as, but not limited to, NovoSeven, fresh frozen plasma, vitamin K, Kcentra or Feiba)
11. Untreatable elevated activated partial thromboplastin time (aPTT)
12. Patients with a mechanical heart valve (presence of bioprosthetic valve(s) is permitted)
13. Positive urine or serum pregnancy test in female subjects without documented history of surgical sterilization or is post-menopausal
14. Participation in a concurrent interventional medical investigation or clinical trial
15. Known life-expectancy of less than 6 months, no reasonable expectation of recovery, Do-Not-Resuscitate (DNR), or comfort measures only prior to randomization
16. Inability or unwillingness of subject or legal guardian/representative to give written informed consent
17. Homelessness or history of drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
18. intolerance or allergy to any TZD1
19. T2DM treated with insulin or an oral medication including Glyburide, unless the NICU physician deems it safe to replace the T2DM medication with pioglitazone1
20. heart failure (symptomatic or NYHA Class I-IV or newly diagnosed on admission TTE screening)
21. patients with abnormal (>1x upper limit of normal) of alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Functional Improvement - modified Rankin Scale (mRS) | 180 Days
  Functional Improvement as determined by utility-weighted modified Rankin Scale (mRS) at 180 days. This is a scale from 0 to 6, where 0 is the best score (no symptoms) and 6 is the worst score.

SECONDARY OUTCOMES:
Efficacy as demonstrated by hematoma clearance | 7 Days
  Determination whether there is non-inferiority or a trend toward more rapid hematoma clearance and perihematomal edema in Group 1 compared to the control arm (Group 2) as measured by serial CT scans during hospitalization residual clot on CT, perihematomal edema on CT
Safety: Number of Participants with 30-day mortality | 30 days
  30-day mortality (30 days from intervention)
Safety: hemorrhage volume | 24 Hours
  increase in hemorrhage volume between index CT and 24-hour follow-up CT
Safety: Number of Participants with bacterial brain infection | 30 Days
  30-day bacterial brain infection (30 days from intervention)
Safety: Number of Participants with hypoglycemia | 30, 90, 120, and 180 days
  occurrences of Moderate hypoglycemia (<70 mg/dL) or Severe hypoglycemia (<50 mg/dL) requiring rescue therapy
Safety: Number of Participants with Drug Toxicity | 30, 90, 120, and 180 days
Economic | 30, 90, 120, and 180 days
  Economic differential as determined by quantification of the cost per quality-adjusted life-years (QALY). QALY uses a scale of 0.00 (dead) to 1.00 (perfect health) for each health status. It is the product of duration of life and a measurement of quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States